CLINICAL TRIAL: NCT04159675
Title: Effect of Burosumab and 1-25 (OH) Vitamin D on Human Osteoblasts From Patients Requiring Craniosynostosis Surgery for Idiopathic Reason or Due to Hypophosphatemic Rickets (HR)
Brief Title: Burosumab and 1-25 (OH) Vitamin D on Human Osteoblasts
Acronym: HYPO-BLASTES
Status: Recruiting | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL19_0773; 2019-A02762-55 (Other: ID-RCB)
Record Dates: First submitted 2019-11-07; First posted 2019-11-12 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Craniosynostoses
MeSH Terms: conditions — Craniosynostoses

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — pieces of bone skull (considered as biological waste) during surgery
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- control patients: Patients with idiopathic craniosynostosis
  Interventions: Biological: osteoblast biology study
- HR patients: Patients with craniosynostosis due to HR
  Interventions: Biological: osteoblast biology study

INTERVENTIONS:
Biological: osteoblast biology study — Describe the in-vitro action of burosumab and vitamin D on human osteoblastogenesis from osteoblasts from patients with craniosynostosis due to HR

SUMMARY:
FGF23 is the cornerstone of phosphate / calcium / vitamin D metabolism: it is synthesized mainly by osteocytes and acts as a phosphaturizing agent, inhibitor of dihydroxyvitamin D, and inhibitor of synthesis and secretion of PTH in most tissues.

The specific role of FGF23 on bone has yet to be demonstrated. In osteoblasts, overexpression of FGF23 in vitro suppresses not only osteoblastic differentiation but also the synthesis of the mineralized matrix independently of its systemic action on phosphate metabolism. In osteoblasts, FGF23 also regulates the secretion of osteopontin by directly suppressing transcription of alkaline phosphatase.

In some diseases such as hypophosphatemic rickets (HR), the direct role of FGF23 on bone has not yet been studied to our knowledge, whereas these genetic hypophosphatemias are secondary to overexpression of FGF23, whether an activating mutation of FGF23 or inhibitory mutations of its inhibitors (DMP1 and PHEX). However, patients with X-linked hypophosphatemic rickets (XLH) have higher circulating FGF23 levels than healthy controls and these levels are higher in treated patients.

Management of XLH consists primarily of correcting the native vitamin D defect by prescribing active vitamin D analogs as well as phosphate supplementation to improve bone mineralization and decrease dental complications, growth, and bone deformities. Recently, a new therapeutic option has been developed for XLH, burosumab, a human monoclonal antibody that binds and inhibits FGF23 activity. The use of burosumab is currently authorized in France in some pediatric patients with severe forms of XLH.

Independently of the indirect bone effects of phosphate correction and vitamin D levels, the direct role of burosumab on bone cells has never been studied. The objective of this project is to study the osteoblastic biology of patients with RH compared to control patients, and to evaluate the direct impact of the treatments used in this pathology on human osteoblasts.

ELIGIBILITY:
Inclusion Criteria:

* Children from 4 months-old to 18 years-old
* Patients requiring craniosynostosis surgery followed by reference centers for rare diseases of calcium and phosphate metabolism / craniofacial malformations
* Patients and parent / holder of parental authority who have been informed of the study and do not object to participate

Exclusion Criteria:

* Patient being treated with oral corticosteroid or having received more than 3 months of corticosteroid treatment before surgery.

Ages: 4 Months to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: patients with craniosynostosis, idiopathic (control patients) or due to HR
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2020-09-04 (Actual); Primary Completion 2026-04-04 (Estimated); Study Completion 2026-04-04 (Estimated)

PRIMARY OUTCOMES:
Number of osteoblastic cells obtained at the end of differentiation | Day 0
  The analysis of osteoblastic differentiation obtained from the bone cells from patients with burosumab and/or 1-25 (OH) vitamin D (HR patients vs idiopathic craniosynostosis)

CONTACTS AND LOCATIONS:
Overall Officials: Federico DI ROCCO, MD, Principal Investigator — Hospices Civils de Lyon Centre de référence des craniosténoses et malformations cranio-faciales Service de neurochirurgie Pédiatrique
Locations (1):
- Centre de référence des craniosténoses et malformations cranio-faciales Service de neurochirurgie Pédiatrique, Bron, France